CLINICAL TRIAL: NCT02565745
Title: Impact of Skin Dressings Compared With Cream for Skin Lubrication in the Prevention of Pressure Ulcers in Patients at High or Very High Risk: A Multicenter Randomized Trial
Brief Title: Skin Dressings Versus Lubrication to Prevent Pressure Ulcers: A Randomized Trial
Acronym: PENFUP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recommendation after interim analysis
Sponsor: Fundación Cardioinfantil Instituto de Cardiología (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2222-2015; 277865740699 (Other Grant/Funding Number: Colciencias)
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2017-06

CONDITIONS: Pressure Ulcer
Keywords: Prevention; Pressure ulcers; Clinical trial; Nursing
MeSH Terms: conditions — Pressure Ulcer | interventions — Biological Dressings; Bandages, Hydrocolloid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors unaware of the treatment allocation will be sent photographs of the target skin areas with suspected PUs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin Dressing (Experimental): Hydrocolloid dressings applied during hospitalization
  Interventions: Combination Product: Skin dressing
- Moisturizing cream (Active Comparator): Use of moisturizing cream, as part of conventional skin care
  Interventions: Other: Moisturizing cream

INTERVENTIONS:
Combination Product: Skin dressing — Pre-determined skin areas at risk for PUs (3 or more, depending on the prevaliing body position, prone, supine or Sims') will be covered. Dressings will be changed every 6-7 days unless found wet/contaminated
  Other Names: Hydrocolloid dressing
  Arms: Skin Dressing
Other: Moisturizing cream — It will be applied twice a day to the same skin areas as the experimental group
  Other Names: Skin lubricant
  Arms: Moisturizing cream

SUMMARY:
Study purpose:

To assess if - in adult patients admitted to hospital with surgical or medical conditions at high/very high risk of developing pressure ulcers (PU) according to Braden scale - using skin dressing protection versus conventional care (lubricant or moisturizer cream) may prevent the incidence of in-hospital PU

DETAILED DESCRIPTION:
Participants will receive, in addition to the experimental/control interventions, background skin care measures, including anti- bedsore mattresses; body position changes every two hours, and shear/friction reduction.

Trained nurses will review all participants' charts and verify any report of PU until the first ambulation, discharge or death. Patients with a verified PU are referred to the institutional wound care group.

For the purpose of outcome adjudication, study personnel will email digital pictures to 2 independent, blinded outcome assessors (experts in skin care). Skin lesions will be rated in 4-level scale (EPUAP/NPUAP). In case of disagreement, a single, independent referee will confirm the presence/absence of any potential PU.

The unit for analysis will be patients developing (first occurrence, in a time-to-event analysis) PUs in the areas covered by the interventions.

See further details on eligibility, interventions and study outcomes below

ELIGIBILITY:
Inpatients will be eligible if meeting two criteria:

* Intact skin on hospital admission
* High/very high risk of PU (Braden´s scale ≤ 20 points) will be eligible.

Exclusion Criteria:

* Treating physician disagree with participation
* Need for chronic use of diapers

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 689 (Actual)
Dates: Start 2015-12; Primary Completion 2017-08-31 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Pressure ulcers | During hospitalization
  First skin ulcer identified in the covered body areas

SECONDARY OUTCOMES:
Length of stay | During hospitalization
  Total stay in hours
Time to the first walk | During hospitalization
  First walk out of bed as registered in patients' charts
Total cost of hospitalization | During hospitalization
  Total bill to insurer

CONTACTS AND LOCATIONS:
Overall Officials: Olga L Cortés, RN,MSC,PhD, Principal Investigator — Fundacion Cardioinfantil Instituto de Cardiología
Locations (2):
- Colombia (2):
  - Fundación Cardioinfantil Instituto de Cardiología, Bogotá, Cundinamarca
  - Clinica Carlos Ardila Lulle-FOSCAL, Bucaramanga, Santander Department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bergstrom N, Allman RM, Alvarez OM, Bennett MA, Carlson CE, Frantz RA, Garber SL, Jackson BS, Kaminski Jr MV, Kemp MG, Krouskop TA, Lewis Jr VL, Maklebust J, Margolis DJ, Marvel EM, Reger SI, Rodeheaver GT, Salcido R, Xakellis GC, Yarkony GM. Treatment of pressure ulcers. Clinical Practice Guideline, No. 15. 1994. AHCPR Publication No. 95-0652. Rockville, MD: U.S. Bergstrom, N, Braden, B, Champagne, M, Kemp, M, & Ruby, E. Predicting pressure ulcer risk: a multisite study of the predictive validity of the Braden Scale. Nursing Research, 1998;47(5):261-269.
- [Result] Moore ZE, Webster J. Dressings and topical agents for preventing pressure ulcers. Cochrane Database Syst Rev. 2013 Aug 18;(8):CD009362. doi: 10.1002/14651858.CD009362.pub2. PMID 23955535
- [Result] McInnes E, Jammali-Blasi A, Bell-Syer SE, Dumville JC, Cullum N. Support surfaces for pressure ulcer prevention. Cochrane Database Syst Rev. 2011 Apr 13;(4):CD001735. doi: 10.1002/14651858.CD001735.pub4. PMID 21491384
- [Derived] Cortes OL, Herrera VM, Salazar LD, Rojas YA, Esparza M, Taborda A, Dennis RJ. Impact of hydrocolloid dressings in the prevention of pressure ulcers in high-risk patients: a randomized controlled trial (PENFUP). Sci Rep. 2023 Dec 7;13(1):21639. doi: 10.1038/s41598-023-47483-0. PMID 38062132